CLINICAL TRIAL: NCT03228082
Title: Blood Pressure After PREeclampsia/HELLP by SELF Monitoring
Brief Title: Blood Pressure After PREeclampsia/HELLP by SELF Monitoring Study
Acronym: BP-PRESELF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Collaborators: Interreg (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Device Feasibility
Other Study IDs: NL59836.091.16
Record Dates: First submitted 2017-06-15; First posted 2017-07-24 (Actual); Last update posted 2020-10-06 (Actual); Status verified 2020-10

CONDITIONS: Preeclampsia; Cardiovascular Risk Factor; Cardiovascular Diseases; Hypertension
Keywords: Patient empowerment; Women's Health; Home Blood Pressure Monitoring
MeSH Terms: conditions — Pre-Eclampsia; Cardiovascular Diseases; Hypertension; Patient Participation | interventions — Blood Pressure Monitoring, Ambulatory

STUDY DESIGN:
Intervention Model Description: Participants will be randomized at the end of the baseline visit to self-measurement of bloodpressure at home (intervention group) or usual care (control group).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Home Blood Pressure Monitoring (HBPM) (Experimental): Home monitoring of blood pressure will be performed. Blood pressure measurements will be entered automatically through a smartphone application into a patient-controlled medical record ('Patients Know Best'). The data will be available to the study coordinator, who will provide patients within 1 week with feedback on the measurements. If necessary lifestyle advice will be given, in case of hypertension patients will be referred to their GP.
  Once monthly a questionnaire on well-being (SF-12) and symptoms will be completed. After 6 months and 1 year patients will also receive a questionnaire on feasibility and usability of the blood pressure device.
  Interventions: Device: Home Blood Pressure Monitoring (HBPM)
- Control group (No Intervention): Patients in the control group will be asked to register their blood pressure if measured during a doctor's visit, and to note medication use if applicable. They will also be asked to complete a short questionnaire on well-being (SF-12) once per month, which will be evaluated at the end of the study. No interim contact with the study coordinator is scheduled.

INTERVENTIONS:
Device: Home Blood Pressure Monitoring (HBPM) — Home blood pressure monitoring using the Withings Wireless BP monitor. Patients will be asked to measure their blood pressure twice daily for 7 consecutive days. This will be repeated for every month for 1 year.
  Arms: Home Blood Pressure Monitoring (HBPM)

SUMMARY:
RATIONALE:

Women with a previous history of preeclampsia (PE)/HELLP have a twofold higher risk of cardiovascular disease (CVD) and a fourfold increased risk to develop hypertension at a relative young age. In the latest 2016 ESC guidelines 'CVD prevention', previous PE has been acknowledged as a serious CVD risk factor in women. In clinical practice, however, these women are still underappreciated for their CVD risk. It has not been established yet how adequate lifelong prevention in these potentially high risk women can optimally be achieved from their childbearing years onwards.

OBJECTIVE:

To evaluate feasibility, usability, acceptance and potential obstacles of blood pressure (BP) home monitoring in high-risk women, aged 40-60 years, after a previous PE in pregnancy. In addition to evaluate the effectiveness of BP home monitoring on the occurrence of hypertension, the efficacy of BP treatment, quality of life (QOL), health-related symptoms, work ability and life-style behaviour.

STUDY DESIGN:

Randomized, open label feasibility study to compare eHealth guided self management of BP monitoring and lifestyle advice with 'usual care'.

STUDY POPULATION:

Approximately 200 women, aged ≥ 40 and ≤ 60 years, with a previous PE in pregnancy will be invited to participate (both early and late PE). Patients will be recruited from the departments of obstetrics/gynaecology in 6 centres in the Euregio Rhein-Waal and from the department of cardiology Radboudumc.

INTERVENTION:

eHealth guided measurements of BP at regular intervals and recurrent lifestyle advice (intervention-group) will be compared with "usual care".

PRIMARY OUTCOME:

Feasibility, usability, acceptance and potential obstacles of BP home monitoring in high-risk women after a previous PE in pregnancy at 1 year of follow-up.

ELIGIBILITY:
Inclusion Criteria:

* previous preeclampsia/HELLP syndrome, defined as diastolic BP≥90 mmHg with proteinuria ≥ 0.3gram/24 h, during one or more pregnancies, more than 1 year ago.
* 'early' or 'late' PE/HELLP
* age ≥40 and ≤ 60 years

Exclusion Criteria:

* pregnant women or women wishing for future pregnancie(s)
* inability to perform self BP measurements
* not having a smartphone (Apple or Android)
* already having regular hypertension control by GP or medical specialist
* previous cardiovascular events, such as myocardial infarction , stroke, heart failure and symptomatic ischemic heart disease

Ages: 40 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 200 (Actual)
Dates: Start 2017-07-13 (Actual); Primary Completion 2019-12-30 (Actual); Study Completion 2019-12-30 (Actual)

PRIMARY OUTCOMES:
Feasibility of HBPM after a previous preeclampsia to evaluate the prevalence of hypertension. | 1 year
  To evaluate feasibility of blood pressure home monitoring to diagnose hypertension at 1 year follow-up, in high-risk women with a previous preeclampsia. Feasibility will be measured using questionnaires (Likert scales).

SECONDARY OUTCOMES:
Blood pressure values | 1 year
  Mean BP values (mmHg) in both study groups at 1 year of follow-up
Prevalence of hypertension | 1 year
  Prevalence of hypertension in both groups at 1 year of follow-up
Effect HBPM | 1 year
  Effect of regular self measurements on blood pressure levels at home at 1 year follow-up

OTHER OUTCOMES:
Quality of Life | 1 year
  QOL measures related to blood pressure by repeated validated questionnaires
Occupational activity | 1 year
  Questionnaires on ability to work and work-related obstacles
BP patterns | 1 year
  Patterns of BP levels and incidence of hypertension during follow-up
Cardiac symptoms | 1 year
  Cardiac symptoms and blood-pressure related symptoms
Costs | 1 year
  Cost-effectiveness of BP self-management versus regular office-based visits

CONTACTS AND LOCATIONS:
Overall Officials: A.H.E.M. Maas, Prof.dr., Principal Investigator — Radboudumc, department Cardiology
Locations (6):
- Germany (3):
  - Katholisches Karl-Leisner-Klinikum GmbH, Kleve
  - Krankenhaus Bethanien, Moers
  - St. Josef Krankenhaus GmbH, Moers
- Netherlands (3):
  - Rijnstate Ziekenhuis, Arnhem
  - Radboudumc, Nijmegen
  - Canisius-Wilhelmina Ziekenhuis, Nijmegen

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Arrieta A, Woods JR, Qiao N, Jay SJ. Cost-benefit analysis of home blood pressure monitoring in hypertension diagnosis and treatment: an insurer perspective. Hypertension. 2014 Oct;64(4):891-6. doi: 10.1161/HYPERTENSIONAHA.114.03780. Epub 2014 Jul 14. PMID 25024284
- [Background] Bellamy L, Casas JP, Hingorani AD, Williams DJ. Pre-eclampsia and risk of cardiovascular disease and cancer in later life: systematic review and meta-analysis. BMJ. 2007 Nov 10;335(7627):974. doi: 10.1136/bmj.39335.385301.BE. Epub 2007 Nov 1. PMID 17975258
- [Background] Brown MC, Best KE, Pearce MS, Waugh J, Robson SC, Bell R. Cardiovascular disease risk in women with pre-eclampsia: systematic review and meta-analysis. Eur J Epidemiol. 2013 Jan;28(1):1-19. doi: 10.1007/s10654-013-9762-6. Epub 2013 Feb 9. PMID 23397514
- [Background] Bushnell C, McCullough LD, Awad IA, Chireau MV, Fedder WN, Furie KL, Howard VJ, Lichtman JH, Lisabeth LD, Pina IL, Reeves MJ, Rexrode KM, Saposnik G, Singh V, Towfighi A, Vaccarino V, Walters MR; American Heart Association Stroke Council; Council on Cardiovascular and Stroke Nursing; Council on Clinical Cardiology; Council on Epidemiology and Prevention; Council for High Blood Pressure Research. Guidelines for the prevention of stroke in women: a statement for healthcare professionals from the American Heart Association/American Stroke Association. Stroke. 2014 May;45(5):1545-88. doi: 10.1161/01.str.0000442009.06663.48. Epub 2014 Feb 6. PMID 24503673
- [Background] Drost JT, Arpaci G, Ottervanger JP, de Boer MJ, van Eyck J, van der Schouw YT, Maas AH. Cardiovascular risk factors in women 10 years post early preeclampsia: the Preeclampsia Risk EValuation in FEMales study (PREVFEM). Eur J Prev Cardiol. 2012 Oct;19(5):1138-44. doi: 10.1177/1741826711421079. Epub 2011 Aug 22. PMID 21859777
- [Background] Heida KY, Bots ML, de Groot CJ, van Dunne FM, Hammoud NM, Hoek A, Laven JS, Maas AH, Roeters van Lennep JE, Velthuis BK, Franx A. Cardiovascular risk management after reproductive and pregnancy-related disorders: A Dutch multidisciplinary evidence-based guideline. Eur J Prev Cardiol. 2016 Nov;23(17):1863-1879. doi: 10.1177/2047487316659573. Epub 2016 Jul 18. PMID 27432836
- [Background] ESH/ESC Task Force for the Management of Arterial Hypertension. 2013 Practice guidelines for the management of arterial hypertension of the European Society of Hypertension (ESH) and the European Society of Cardiology (ESC): ESH/ESC Task Force for the Management of Arterial Hypertension. J Hypertens. 2013 Oct;31(10):1925-38. doi: 10.1097/HJH.0b013e328364ca4c. No abstract available. PMID 24107724
- [Background] Mannisto T, Mendola P, Vaarasmaki M, Jarvelin MR, Hartikainen AL, Pouta A, Suvanto E. Elevated blood pressure in pregnancy and subsequent chronic disease risk. Circulation. 2013 Feb 12;127(6):681-90. doi: 10.1161/CIRCULATIONAHA.112.128751. PMID 23401113
- [Background] Margolis KL, Asche SE, Bergdall AR, Dehmer SP, Groen SE, Kadrmas HM, Kerby TJ, Klotzle KJ, Maciosek MV, Michels RD, O'Connor PJ, Pritchard RA, Sekenski JL, Sperl-Hillen JM, Trower NK. Effect of home blood pressure telemonitoring and pharmacist management on blood pressure control: a cluster randomized clinical trial. JAMA. 2013 Jul 3;310(1):46-56. doi: 10.1001/jama.2013.6549. PMID 23821088
- [Background] McDonald SD, Malinowski A, Zhou Q, Yusuf S, Devereaux PJ. Cardiovascular sequelae of preeclampsia/eclampsia: a systematic review and meta-analyses. Am Heart J. 2008 Nov;156(5):918-30. doi: 10.1016/j.ahj.2008.06.042. Epub 2008 Oct 2. PMID 19061708
- [Background] McManus RJ, Mant J, Bray EP, Holder R, Jones MI, Greenfield S, Kaambwa B, Banting M, Bryan S, Little P, Williams B, Hobbs FD. Telemonitoring and self-management in the control of hypertension (TASMINH2): a randomised controlled trial. Lancet. 2010 Jul 17;376(9736):163-72. doi: 10.1016/S0140-6736(10)60964-6. Epub 2010 Jul 8. PMID 20619448
- [Background] McManus RJ, Mant J, Haque MS, Bray EP, Bryan S, Greenfield SM, Jones MI, Jowett S, Little P, Penaloza C, Schwartz C, Shackleford H, Shovelton C, Varghese J, Williams B, Hobbs FD, Gooding T, Morrey I, Fisher C, Buckley D. Effect of self-monitoring and medication self-titration on systolic blood pressure in hypertensive patients at high risk of cardiovascular disease: the TASMIN-SR randomized clinical trial. JAMA. 2014 Aug 27;312(8):799-808. doi: 10.1001/jama.2014.10057. PMID 25157723
- [Background] Mosca L, Benjamin EJ, Berra K, Bezanson JL, Dolor RJ, Lloyd-Jones DM, Newby LK, Pina IL, Roger VL, Shaw LJ, Zhao D, Beckie TM, Bushnell C, D'Armiento J, Kris-Etherton PM, Fang J, Ganiats TG, Gomes AS, Gracia CR, Haan CK, Jackson EA, Judelson DR, Kelepouris E, Lavie CJ, Moore A, Nussmeier NA, Ofili E, Oparil S, Ouyang P, Pinn VW, Sherif K, Smith SC Jr, Sopko G, Chandra-Strobos N, Urbina EM, Vaccarino V, Wenger NK. Effectiveness-based guidelines for the prevention of cardiovascular disease in women--2011 update: a guideline from the american heart association. Circulation. 2011 Mar 22;123(11):1243-62. doi: 10.1161/CIR.0b013e31820faaf8. Epub 2011 Feb 14. No abstract available. PMID 21325087
- [Background] Writing Group Members; Mozaffarian D, Benjamin EJ, Go AS, Arnett DK, Blaha MJ, Cushman M, Das SR, de Ferranti S, Despres JP, Fullerton HJ, Howard VJ, Huffman MD, Isasi CR, Jimenez MC, Judd SE, Kissela BM, Lichtman JH, Lisabeth LD, Liu S, Mackey RH, Magid DJ, McGuire DK, Mohler ER 3rd, Moy CS, Muntner P, Mussolino ME, Nasir K, Neumar RW, Nichol G, Palaniappan L, Pandey DK, Reeves MJ, Rodriguez CJ, Rosamond W, Sorlie PD, Stein J, Towfighi A, Turan TN, Virani SS, Woo D, Yeh RW, Turner MB; American Heart Association Statistics Committee; Stroke Statistics Subcommittee. Heart Disease and Stroke Statistics-2016 Update: A Report From the American Heart Association. Circulation. 2016 Jan 26;133(4):e38-360. doi: 10.1161/CIR.0000000000000350. Epub 2015 Dec 16. No abstract available. PMID 26673558
- [Background] Piepoli MF, Hoes AW, Agewall S, Albus C, Brotons C, Catapano AL, Cooney MT, Corra U, Cosyns B, Deaton C, Graham I, Hall MS, Hobbs FDR, Lochen ML, Lollgen H, Marques-Vidal P, Perk J, Prescott E, Redon J, Richter DJ, Sattar N, Smulders Y, Tiberi M, van der Worp HB, van Dis I, Verschuren WMM, Binno S; ESC Scientific Document Group. 2016 European Guidelines on cardiovascular disease prevention in clinical practice: The Sixth Joint Task Force of the European Society of Cardiology and Other Societies on Cardiovascular Disease Prevention in Clinical Practice (constituted by representatives of 10 societies and by invited experts)Developed with the special contribution of the European Association for Cardiovascular Prevention & Rehabilitation (EACPR). Eur Heart J. 2016 Aug 1;37(29):2315-2381. doi: 10.1093/eurheartj/ehw106. Epub 2016 May 23. No abstract available. PMID 27222591
- [Background] Spaan J, Peeters L, Spaanderman M, Brown M. Cardiovascular risk management after a hypertensive disorder of pregnancy. Hypertension. 2012 Dec;60(6):1368-73. doi: 10.1161/HYPERTENSIONAHA.112.198812. Epub 2012 Oct 15. No abstract available. PMID 23071130
- [Background] Verberk WJ, Kroon AA, Lenders JW, Kessels AG, van Montfrans GA, Smit AJ, van der Kuy PH, Nelemans PJ, Rennenberg RJ, Grobbee DE, Beltman FW, Joore MA, Brunenberg DE, Dirksen C, Thien T, de Leeuw PW; Home Versus Office Measurement, Reduction of Unnecessary Treatment Study Investigators. Self-measurement of blood pressure at home reduces the need for antihypertensive drugs: a randomized, controlled trial. Hypertension. 2007 Dec;50(6):1019-25. doi: 10.1161/HYPERTENSIONAHA.107.094193. Epub 2007 Oct 15. PMID 17938383
- [Derived] Muijsers HEC, van der Heijden OWH, de Boer K, van Bijsterveldt C, Buijs C, Pagels J, Tonnies P, Heiden S, Roeleveld N, Maas AHEM. Blood pressure after PREeclampsia/HELLP by SELF monitoring (BP-PRESELF): rationale and design of a multicenter randomized controlled trial. BMC Womens Health. 2020 Mar 4;20(1):41. doi: 10.1186/s12905-020-00910-0. PMID 32131802